CLINICAL TRIAL: NCT01057615
Title: Comparative and Additive Effects of Fish Oil and Ascorbic Acid Supplementation on Exercise-Induced Bronchoconstriction and Airway Inflammation in Asthma
Brief Title: Effect of Fish Oil and Vitamin C on Exercise-Induced Bronchoconstriction and Airway Inflammation in Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Timothy Mickleborough, PhD / Associate Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0910000751
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Last update posted 2011-01-31 (Estimated); Status verified 2011-01

CONDITIONS: Asthma
Keywords: Asthma; Exercise-Induced Bronchoconstriction; Inflammation; Airway; Fish Oil; Ascorbic Acid
MeSH Terms: conditions — Asthma; Inflammation | interventions — Fish Oils; Ascorbic Acid; Soybean Oil; Dietary Sucrose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Active Fish Oil + Vitamin C Placebo (Experimental): Fifteen subjects will take 10 active fish oil capsules per day and 2 vitamin C placebo capsules per day for 3 weeks.
  Interventions: Dietary Supplement: Fish Oil; Dietary Supplement: Ascorbic Acid Placebo
- Fish Oil Placebo + Active Vitamin C (Experimental): Fifteen subjects will take 10 fish oil placebo capsules per day and 2 active vitamin C capsules per day for 3 weeks.
  Interventions: Dietary Supplement: Ascorbic Acid; Dietary Supplement: Fish Oil Placebo
- Active Fish Oil + Active Vitamin C (Experimental): Following a 2-week washout period, all subjects from the other two arms (n=30) will take 10 active fish oil capsules per day and 2 active vitamin C capsules per day for 3 weeks.
  Interventions: Dietary Supplement: Fish Oil; Dietary Supplement: Ascorbic Acid

INTERVENTIONS:
Dietary Supplement: Fish Oil — 10 fish oil (3.2g EPA + 2.0g DHA) capsules per day for 3 weeks
  Arms: Active Fish Oil + Active Vitamin C; Active Fish Oil + Vitamin C Placebo
Dietary Supplement: Ascorbic Acid — 2 pharmaceutical grade ascorbic acid (1500mg) capsules per day for 3 weeks
  Other Names: Vitamin C
  Arms: Active Fish Oil + Active Vitamin C; Fish Oil Placebo + Active Vitamin C
Dietary Supplement: Fish Oil Placebo — 10 placebo fish oil (soy bean oil) capsules per day for 3 weeks
  Other Names: Soy Bean Oil
  Arms: Fish Oil Placebo + Active Vitamin C
Dietary Supplement: Ascorbic Acid Placebo — 2 placebo ascorbic acid (sucrose) capsules per day for 3 weeks
  Other Names: Table Sugar
  Arms: Active Fish Oil + Vitamin C Placebo

SUMMARY:
Combining fish oil and vitamin C supplementation will provide a greater anti-inflammatory effect against developing exercise-induced bronchoconstriction (EIB) than either nutritional supplement alone.

DETAILED DESCRIPTION:
The aim of this study is to extend previous findings that nutritional supplementation or dietary modification can ameliorate exercise-induced bronchoconstriction. It has been shown in separate studies that fish oil and ascorbic acid (vitamin C) individually protect against EIB by improving pulmonary function and reducing airway inflammation. The main aim of this study is to determine the comparative and additive effects of fish oil and ascorbic acid supplementation on EIB and airway inflammation in asthmatic individuals.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma, based on medication use as well as history and symptoms as outlined in the NHLBI Guidelines for the Diagnosis and Management of Asthma
* Diagnosis of EIB, based on ≥10% fall in post-challenge FEV1, a measure of lung function, after dry air eucapnic voluntary hyperventilation (EVH), a simulated exercise challenge
* Not currently taking asthma maintenance medication or physician approval to discontinue current asthma medication for the duration of the study
* Not currently taking any fish oil or ascorbic acid supplements above the level recommended for adequate intake (if currently taking supplements, can participate if the subject stops taking the supplements for 2 weeks before starting the study and throughout the study)
* Agree to limit fish consumption to 1 fish meal per week throughout the study
* Agree to avoid vitamin C-rich foods throughout the study

Exclusion Criteria:

* Resting FEV1 (the amount of air blown out in the first second of a forced exhalation) <60% of predicted when off medication
* Pregnancy
* History of cardiovascular disease, including hyperlipidemia (high cholesterol) and hypertension (high blood pressure)
* History of bleeding disorders or delayed clotting time
* History of diabetes
* History of seizures
* Allergy to fish oil or ascorbic acid (vitamin C)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2010-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Pulmonary Function | 8 weeks

SECONDARY OUTCOMES:
Exhaled nitric oxide to measure airway inflammation | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Timothy D Mickleborough, PhD, Study Director — Indiana University
Locations (1):
- Indiana University, Bloomington, Indiana, United States

REFERENCES:
- [Background] Mickleborough TD, Murray RL, Ionescu AA, Lindley MR. Fish oil supplementation reduces severity of exercise-induced bronchoconstriction in elite athletes. Am J Respir Crit Care Med. 2003 Nov 15;168(10):1181-9. doi: 10.1164/rccm.200303-373OC. Epub 2003 Aug 6. PMID 12904324
- [Background] Mickleborough TD, Lindley MR, Ionescu AA, Fly AD. Protective effect of fish oil supplementation on exercise-induced bronchoconstriction in asthma. Chest. 2006 Jan;129(1):39-49. doi: 10.1378/chest.129.1.39. PMID 16424411
- [Background] Tecklenburg SL, Mickleborough TD, Fly AD, Bai Y, Stager JM. Ascorbic acid supplementation attenuates exercise-induced bronchoconstriction in patients with asthma. Respir Med. 2007 Aug;101(8):1770-8. doi: 10.1016/j.rmed.2007.02.014. Epub 2007 Apr 5. PMID 17412579